CLINICAL TRIAL: NCT02964429
Title: Determination of the In-vivo Ultrafiltration Coefficient and Evaluation of Performance, Hemo- and Biocompatibility- and Safety-data of High Flux Hemodialyser Diacap Pro in Patients With End Stage Renal Disease on Chronic Hemodialysis
Brief Title: Determination In-vivo KUF for Diacap Pro Hemodialyser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.Braun Avitum AG (Industry)
Collaborators: Winicker Norimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BA-G-H-1602
Record Dates: First submitted 2016-10-28; First posted 2016-11-16 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Kidney Failure,Chronic; Renal Insufficiency,Chronic; Kidney Disease, End-Stage; Kidney Insufficiency
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diacap Pro High-Flux (Experimental): 1.3/ 1.6/ 1.9 sqm
  Interventions: Device: Diacap Pro High-Flux

INTERVENTIONS:
Device: Diacap Pro High-Flux — During dialysis treatment ultrafiltration rate will be changed following a fixed schedule and resulting changes in Transmembrane Pressure (TMP) recorded to generate data for calculation of the in-vivo KUF.

SUMMARY:
The main purpose of this study is the determination of the in-vivo ultrafiltration coefficient (in-vivo KUF) for Diacap Pro dialyzers following routine dialysis prescription in the United States.

DETAILED DESCRIPTION:
The in-vivo KUF for Diacap Pro High Flux dialysers with the surface sizes of 1.3/ 1.6/ 1.9 sqm will be determined as required by the US guideline "Guidance for the Content of Premarket Notifications for Conventional and High Permeability Hemodialyzers 1998" for comparison with the in-vitro KUF data.

Clinical data of at least 12 patients will be collected for determination of the in-vivo KUF complemented by safety-, performance-data for the removal of small and middle molecular substances and hemocompatibility data.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from patient or parents/ guardian.
2. Subject age > 18
3. Effective blood flow 350 ml/min and dialysate flow in the range of 500 - 800 ml/min
4. On hemodialysis for a minimum of 3 months
5. Use of Cimino- or Gore-tex shunts
6. Routine dialysis-treatment for 240 min and 3 times per week
7. Documented dialysis adequacy parameter spKt/V >=1.2 that has been stable for past 3 months
8. Plan to dialyze at participating hemodialysis center for at least 3-months duration.
9. Free from any currently known unusual clotting or access problems
10. Hepatitis B surface antigen (HbsAg) negative, documented within the past 90 days or Hepatitis B surface antibody (anti-HBs) positive.
11. Anti HCV negative, documented within the past 90 days
12. Anti HIV negative, documented within the past 90 days Hematocrit (HCT) between 25 and 40% or haemoglobin (Hb) not less than 8 g/dL

Exclusion Criteria:

1. Patients who are unable to tolerate an effective blood flow of 350 ml/min
2. Patients using catheter for dialysis
3. Pregnant or nursing woman. Women of childbearing potential must agree to avoid pregnancy during the study period
4. Previous plan for extended absences from the participating hemodialysis centre
5. Expected to be transplanted (living related donor) within the maximum of 3 months for the study period
6. Any serious medical conditions or disability, which in the opinion of the investigator, would interfere with treatment or assessment or preclude completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
Changes in Transmembrane Pressure (TMP) dependent on differerent ultrafiltration rates for calculation of the in-vivo ultrafiltration coefficient (in-vivo KUF) | For two of three dialysis sessions each week for a total study period of six weeks
  UF-rates will be changed over a range starting from 600 ml/min to 1000 ml/min to 1400 ml/min to finally 1800 ml/min and resulting changes in Transmembrane Pressure (TMP) will be documented.

SECONDARY OUTCOMES:
Clearance data dialyzer [ml/min] | For one of six dialysis sessions each two weeks for a total study period of six weeks
  For ß2M; Myoglobin; Retinol-Binding-Protein; alpha-1-Microglobulin; Albumin clearance data will be assessed by using serum samples pre- and post dialyzer at timepoints t=0 and t=240 min.
Reduction rates dialyzer [%] | For two of three dialysis sessions each week for a total study period of six weeks
  For urea; creatinine; phosphate; ß2-Microglobulin; Myoglobin; Retinol-Binding-Protein; alpha-1 Microglobulin and Albumin reduction rates will be calculated by using serum-levels at timepoints t=0 and t=240 min.
Total removal of proteins [mg/session] | For one of six dialysis sessions each two weeks for a total study period of six weeks
  Spent dialysate will be collected during the entire dialysis treatment. Considering dialysate flow rate and ultrafiltration volume concentration of ß2-Microglobulin; Myoglobin; Retinol-Binding-Protein;alpha-1 Microglobulin; Albumin; Total Protein will be used to calculate total removal by multiplying with the effective spent dialysate volume
Complement-activation C3a and C5a [ng/ml] | For one of six dialysis sessions each two weeks for a total study period of six weeks
  For complement activation C3a [ng/ml]; C5a [ng/ml] will be assessed at timepoints t=0, t=15; t=60; t=240 min.
Complement-activation TAT III [µg/l] | For one of six dialysis sessions each two weeks for a total study period of six weeks
  For complement activation TAT III [µg/l] will be assessed at timepoints t=0, t=15; t=60; t=240 min.
Inflammatory response Interleukin-1, Interleukin-6 and TNF-alpha [pg/ml] | For one of six dialysis sessions each two weeks for a total study period of six weeks
  For inflammatory response Interleukin-1 [pg/ml]; Interleukin-6 [pg/ml]; TNF-alpha will be assessed at timepoints t=0; t=15; t=60; t=240 min
Inflammatory response CRP [mg/l] | For one of six dialysis sessions each two weeks for a total study period of six weeks
  For inflammatory response CRP[mg/l] will be assessed at timepoints t=0; t=15; t=60; t=240 min
Incidence of Treatment-Emergent Adverse Events | November 2016 up to 2 months
  Number of patients presenting adverse events will be assessed following CTCAE v4.0 grading.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Polakovic, Prim. MUDr., Principal Investigator — Interni oddeleni Strahov VFN
Locations (1):
- Interní oddělení Strahov VFN, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No